CLINICAL TRIAL: NCT01085318
Title: A Twenty-four Week, Two Arm, Pilot Trial to Evaluate Remyelination/ Demyelination, Gray Matter Volume and Iron Deposition in the Central Nervous System (CNS) and Immune Status of Subjects With Relapsing-remitting Multiple Sclerosis (RRMS) Treated With Rebif® 44 mcg Subcutaneously (sc) Three Times a Week (Tiw) Compared to a Healthy Control Group
Brief Title: Rebif Advanced Magnetic Resonance Imaging (MRI) and Immunology Pilot Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 29665
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

ARMS (2):
- Arm 1 MS Patients (Active Comparator): Rebif 44 tiw
  Interventions: Drug: Rebif
- Arm 2 Healthy Control (No Intervention)

INTERVENTIONS:
Drug: Rebif — 44 mcg tiw
  Arms: Arm 1 MS Patients

SUMMARY:
The purpose of this trial is to evaluate the effects of Rebif® 44 mcg subcutaneous (sc) three times a week (tiw) on a) remyelination/demyelination, b) lesion and brain volume, c) central nervous system (CNS) iron deposition, and d) immune status in subjects with relapsing-remitting multiple sclerosis (RRMS) RRMS via several MRI techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, 18-65 years of age, inclusive, at the time of informed consent signature
2. RRMS diagnosed according to the McDonald criteria, treatment naïve or currently using any of the FDA-approved DMDs (excluding natalizumab (Tysabri®), mitoxantrone or Rebif®)
3. Have a disease duration of up to twenty years
4. Be willing and able to comply with the study procedures for the duration of the trial
5. Have given written informed consent and signed Health Insurance Portability and Accountability Act (HIPAA) Authorization before any study- related activities are carried out
6. Female subjects must not be either pregnant or breast-feeding and must lack childbearing potential, as defined by either:

The following inclusion criteria must be fulfilled by the Healthy Control subjects:

1. Male and female subjects, 18-65 years of age, inclusive, at the time of informed consent signature
2. Be willing and able to comply with the study procedures for the duration of the trial
3. Have given written informed consent and signed Health Insurance Portability and Accountability Act (HIPAA) Authorization before any study- related activities are carried out
4. Female subjects must not be either pregnant or breast-feeding and must lack childbearing potential, as defined by either:

Exclusion Criteria:

1. Have received treatment within three months prior to Screening with interferon-beta-1a (Rebif®), IVIG or plasmapheresis
2. Have received treatment within thirty days prior to screening with immunosuppressant agents (e.g. including but not limited to mitoxantrone, cyclophosphamide, cladribine, fludarabine, cyclosporine or total body irradiation) or any other concomitant immunomodulatory therapies (e.g., azathioprine, methotrexate, CellCept®, natalizumab, alemtuzumab/Campath and other immunomodulators/monoclonal agents)
3. Have had a relapse within thirty days prior to the Screening Visit
4. Have received steroid treatment within thirty days prior to the initial MRI scan date at Study Day 1
5. Have inadequate liver function, defined by a alanine aminotransferase (ALT) > 2.5x upper limit of normal (ULN), or alkaline phosphatase > 2.5x ULN, or total bilirubin > 1.5x ULN
6. Have inadequate bone marrow reserve, defined as a total white blood cell count < 3.0x 109/L, platelet count < 75x109/L, hemoglobin < 100g/L
7. Have complete transverse myelitis or simultaneous-onset bilateral optic neuritis
8. Have a history of alcohol or drug abuse
9. Have thyroid dysfunction
10. Have moderate to severe renal impairment
11. Have a major medical or psychiatric illness that in the opinion of the investigator creates undue risk to the subject or could affect compliance with the study protocol
12. Have a history of seizures not adequately controlled by treatment
13. Have serious or acute cardiac disease, such as uncontrolled dysrhythmias, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled congestive heart failure
14. Have, in the opinion of the investigator, any visual, physical or cognitive impairment that would preclude the subject from complying with the study protocol
15. Have a known hypersensitivity or allergy to interferon-beta or any of the excipients
16. Have received an investigational drug or experimental procedure within the past thirty days
17. Are pregnant or attempting to conceive

The following exclusion criteria must be fulfilled by the Healthy Control subjects:

1. Have met any of the above noted criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-06-30 (Actual); Primary Completion 2012-02-29 (Actual); Study Completion 2012-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Dangond, MD, Study Director — EMD Serono
Locations (1):
- EMD Serono, Inc., Rockland, Massachusetts, United States

REFERENCES:
- [Result] Dwyer MG, Zivadinov R, Tao Y, Zhang X, Kennedy C, Bergsland N, Ramasamy DP, Durfee J, Hojnacki D, Weinstock-Guttman B, Hayward B, Dangond F, Markovic-Plese S. Immunological and short-term brain volume changes in relapsing forms of multiple sclerosis treated with interferon beta-1a subcutaneously three times weekly: an open-label two-arm trial. BMC Neurol. 2015 Nov 11;15:232. doi: 10.1186/s12883-015-0488-9. PMID 26559139
- [Result] Zivadinov R, Dwyer MG, Markovic-Plese S, Kennedy C, Bergsland N, Ramasamy DP, Durfee J, Hojnacki D, Hayward B, Dangond F, Weinstock-Guttman B. Effect of treatment with interferon beta-1a on changes in voxel-wise magnetization transfer ratio in normal appearing brain tissue and lesions of patients with relapsing-remitting multiple sclerosis: a 24-week, controlled pilot study. PLoS One. 2014 Mar 13;9(3):e91098. doi: 10.1371/journal.pone.0091098. eCollection 2014. PMID 24625687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at the clinic - June 16, 2010 through July 6, 2011
Pre-assignment Details: Relapsing Remitting Multiple Sclerosis (RRMS)Participants could not have received treatment within 3 months prior to Screening with interferon-beta-1a (Rebif®), IVIG or plasmapheresis
Groups:
- Arm 1 RRMS Patients: Rebif 44 mcg sc tiw
- Arm 2 Healthy Control: Healthy Control
Period: Overall Study
Arm/Group | Arm 1 RRMS Patients | Arm 2 Healthy Control
Started | 23 | 15
Completed | 21 | 15
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 RRMS Patients | Arm 2 Healthy Control | Total
Number analyzed (Participants) | 23 | 15 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 15 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (10.17) | 36.7 (10.31) | 38.6 (10.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 23 | 15 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Volume (in Millimeters Cubed) of Normal Appearing Brain Tissue (NABT) With Increasing (Indicative of Remyelination) Voxel-wise Magnetization Transfer Ratio (VW-MTR) From Baseline to 6 Months
Description: To characterize the effect of Rebif on remyelination using VW-MTR dynamic mapping of NABT in subjects ith RRMS over 6 months of treatment compared to a group of healthy Control (HC).
Time Frame: Baseline to Month 6
Population: The analysis were run on the Intent-to-Treat (ITT) set defined as all RRMS subjects with at least one injection of Rebif and all HC who signed the informed consent form. Missing data were not imputed.
Measure: Median (Full Range); unit: mm^3
Arm/Group | Arm 1 RRMS Patients | Arm 2 Healthy Control
Number analyzed (Participants) | 21 | 13
mm^3 | 1206.1 (4081.621) [0 to 15278.1] | 342 (291.890) [0 to 951]
Statistical Analysis 1: Comparison: Arm 1 RRMS Patients vs Arm 2 Healthy Control; Test type: Superiority or Other; p = 0.061, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 864.1

2. Secondary Outcome: Change in Volume (in Millimeters Cubed) of Normal Appearing Brain Tissue (NABT) With Decreasing (Indicative of Demyelination) Voxel-wise Magnetization Transfer Ratio (VW-MTR)From Baseline to 6 Months
Description: To characterize the effect of Rebif on demyelination using VW-MTR dynamic mapping of NABT in subjects ith RRMS over 6 months of treatment compared to a group of healthy Control (HC).
Time Frame: Baseline to Month 6
Measure: Median (Full Range); unit: mm^3
Arm/Group | Arm 1 RRMS Patients | Arm 2 Healthy Control
Number analyzed (Participants) | 21 | 13
mm^3 | 941.99 (1262.565) [0 to 6140.6] | 297 (311.269) [0 to 852]
Statistical Analysis 1: Comparison: Arm 1 RRMS Patients vs Arm 2 Healthy Control; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 644.99

3. Other Pre Specified Outcome: Clinical Relapses
Description: Clinical Relapses
Time Frame: Over 6 months
Measure: Mean (Standard Deviation); unit: relapses per participant
Arm/Group | Arm 1 RRMS Patients
Number analyzed (Participants) | 23
relapses per participant | 0.3 (0.88)

4. Other Pre Specified Outcome: Time to First Clinical Relapse
Description: Time to First Clinical Relapse
Time Frame: Months
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Arm 1 RRMS Patients
Number analyzed (Participants) | 23
months | 2.5 (1.88)

ADVERSE EVENTS:
Arm/Group | Arm 1 RRMS Patients | Arm 2 Healthy Control
Serious Adverse Events (participants affected / at risk) | 2/23 | 0/15
Other Adverse Events (participants affected / at risk) | 22/23 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 RRMS Patients (N=23) | Arm 2 Healthy Control (N=15)
Multiple Sclerosis Relapse (Nervous system disorders) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 RRMS Patients (N=23) | Arm 2 Healthy Control (N=15)
Influenza like illness (General disorders) | 9 | 0
Injection site reaction (General disorders) | 8 | 0
Multiple sclerosis relapse (Nervous system disorders) | 5 | 0
Fatigue (General disorders) | 4 | 0
Injection site pain (General disorders) | 4 | 0
Nasopharyngitis (Infections and infestations) | 4 | 2
Headache (Nervous system disorders) | 3 | 0
Migraine (Nervous system disorders) | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Gastroenteritis viral (Gastrointestinal disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Irritability (General disorders) | 2 | 0
Multiple sclerosis (Nervous system disorders) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither Institution nor any Principal Investigators shall publish or present any results from such Study to any third parties until: (i) EMD Serono publishes the results from all sites participating in such Study; (ii) Institution receives notification from EMD Serono that publication of the multi-site results is no longer planned; or (iii) twenty-four (24) months following the completion of the multi-site study at all sites, whichever occurs first.